CLINICAL TRIAL: NCT06877338
Title: Inspiratory and Trunk Muscle Activity During Inspiratory Muscle Training on Stable and Unstable Surfaces in People After Stroke
Brief Title: Inspiratory and Trunk Muscle Activity During IMT on Stable and Unstable Surfaces in Stroke Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, LIU FANG, PhD student, Hong Kong Metropolitan University
Other Study IDs: No: HE-OT2023/13
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Inspiratory Muscle Training; Diaphragm; Sternocleidomastoid Muscles; Trunk Muscle Activity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Loaded breathing on stable and unstable surfaces — Participants will be instructed to perform 10 loaded breaths via a threshold inspiratory load device on both a stable surface (sitting on a chair, Protocol 1) and an unstable surface (sitting on a soft pad, Protocol 2) in random order. The inspiratory load/resistance will be set at 50% of the maximum inspiratory pressure (MIP).

SUMMARY:
This study aims to investigate the differences in muscle recruitment of the diaphragm (assessed using ultrasound), the sternocleidomastoid (SCM) and trunk muscles (both measured via surface electromyography (sEMG)), during loaded breathing training performed on both stable and unstable surfaces. The goal is to understand the interaction between the inspiratory and trunk muscles during Inspiratory muscle training (IMT) across these two surface conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years and < 80 years
* Breathing spontaneously
* Clinically diagnosed with ischemic and/or hemorrhagic stroke
* Stroke duration from onset between 1 and 12 months
* No thoracic or abdominal surgery in the past 6 months
* No cognitive impairment (Montreal Cognitive Assessment (MoCA) score ≥ 26)
* Able to understand and follow verbal instructions
* No facial palsy or only mild facial palsy without limitation of labial occlusion
* Able to complete all loaded breathing tests on both stable and unstable surfaces included in this study

Exclusion Criteria:

* Acute myocardial infarction or acute heart failure
* Acute pain in any part of the body
* History of chronic respiratory illness or positive clinical signs of impaired respiratory function (such as shortness of breath, hypoxemia, chronic cough, and sputum retention)
* Presence of a nasal feeding tube, tracheal tube, or any condition that prevents the measurement or implementation of the study procedures

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People diagnosed with stroke who meet the criteria will be invited to participate in the study
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | Day 1
  Diaphragmatic thickening fraction is determined by "(thickness of the diaphragm at end inspiratory - thickness at end expiratory)/thickness at end expiratory". Diaphragmatic thickness will be measured by ultrasonography.

SECONDARY OUTCOMES:
Muscle activation of the sternocleidomastoid muscle | Day 1
  Surface electromyography (sEMG) will be used to measure accessory inspiratory muscle (sternocleidomastoid muscles) activity during all breathing protocol tests.
Muscle activation of the trunk muscles | Day 1
  Surface electromyography (sEMG) will be used to measure the muscle activity of rectus abdominis (RA), external oblique (EO), internal oblique/transversus abdominis (IO/TrA), and erector spinae (ES)- using sEMG during all breathing protocol tests.
Perceived Exertion Borg scale | Day 1
  This is a vertical scale quantified from 0 to 10, where 0 represents no symptoms, and 10 represents the maximum symptoms. The Borg score provides an individual measurement of the exercise intensity.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT06877338/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT06877338/ICF_001.pdf